CLINICAL TRIAL: NCT05891639
Title: Investigating Factors Affecting Clinical Trial Participation Rates in Patients With Bipolar Disorder
Brief Title: A Close Examination of Patient Experiences in Bipolar Disorder Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81011326
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in clinical trials usually favors a particular demographic group. But there is limited research available to explain what study attributes affect the completion of these specific demographic groups.

This study will investigate the safety and efficacy of bipolar disorder treatments. The focus will be on tracking the rates of completion and withdrawal among these individuals.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future bipolar disorder study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Diagnosis of bipolar disorder
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Has a serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Inability to perform regular electronic reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are actively considering involvement in an observational bipolar disorder clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of bipolar disorder patients who decide to enroll in a clinical research. | 3 months
Number of bipolar disorder study participants who remain in clinical research until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perugi G, Medda P, Toni C, Mariani MG, Socci C, Mauri M. The Role of Electroconvulsive Therapy (ECT) in Bipolar Disorder: Effectiveness in 522 Patients with Bipolar Depression, Mixed-state, Mania and Catatonic Features. Curr Neuropharmacol. 2017 Apr;15(3):359-371. doi: 10.2174/1570159X14666161017233642. PMID 28503107
- [Background] Yeom JW, Cho CH, Jeon S, Seo JY, Son S, Ahn YM, Kim SJ, Ha TH, Cha B, Moon E, Park DY, Baek JH, Kang HJ, An H, Lee HJ. Bipolar II disorder has the highest prevalence of seasonal affective disorder in early-onset mood disorders: Results from a prospective observational cohort study. Depress Anxiety. 2021 Jun;38(6):661-670. doi: 10.1002/da.23153. Epub 2021 Apr 5. PMID 33818866
- [Background] Rakofsky JJ, Dunlop BW. Treating nonspecific anxiety and anxiety disorders in patients with bipolar disorder: a review. J Clin Psychiatry. 2011 Jan;72(1):81-90. doi: 10.4088/JCP.09r05815gre. Epub 2010 Nov 16. PMID 21208580

DOCUMENTS (1):
  • Informed Consent Form (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT05891639/ICF_000.pdf